CLINICAL TRIAL: NCT06663670
Title: Comparative Effects of Intraneural Facilitation Therapy and Nerve Flossing Technique on Pain, Balance, Gait, and Quality of Life in Patients With Diabetic Peripheral Neuropathy
Brief Title: Intraneural Facilitation Therapy and Nerve Flossing Technique in Patients With Diabetic Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0256
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetes mellitus Type 2; Diabetic Neuropathy; Endoneurium; Epineurium; Gait; Pain; Peripheral Nerve; Quality of Life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as assessor of the study would be kept blind of the treatment groups to which patient will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A Intraneural Facilitation Therapy along with Home care plan (Experimental): Group A will receive 24 sessions of Intraneural Facilitation therapy, delivered three times weekly for eight weeks, each session lasting 60 minutes. Effects will be measured at baseline, post-intervention (after 8 weeks), and at a 2-months follow-up.
  Interventions: Other: Intraneural Facilitation Therapy
- Group B Nerve Flossing Technique along with Home care plan (Experimental): Group B will receive the nerve flossing technique for about 3 sets of 10 repetitions with an interval of 1 minutes between sets. A total of 24 sessions (3x/week for 8 weeks) will be conducted, lasting 50-60 minutes each. The effects will be measured at baseline (pre-treatment), after week 8 (post-intervention), and at 2-month follow-up.
  Interventions: Other: Nerve Flossing Technique

INTERVENTIONS:
Other: Intraneural Facilitation Therapy — * The initial hold, known as the facilitation hold, involves placing the contralateral joint in a maximal loose-pack position that will be comfortable for the patient. An illustration of this would be positioning the ankle joint on the contralateral side in full plantar flexion and inversion. Throughout the entire session, this position will be maintained using a stretch strap. It is crucial to emphasize that there is no muscle engagement in the joint where the facilitation takes place, only a slight stretch.
  * Once the pressure elevation occurs, the subsequent phase known as the secondary hold will be initiated to direct the augmented flow of epineurial blood toward the transperineurial vessels connecting the epiperineum and the endoneurial capillaries of the target area.
  * The final maneuver, the sub hold, leverages Bernoulli's principle to augment blood flow through the ischemic endoneurial capillaries experiencing heightened transmural pressure.
  Arms: GROUP A Intraneural Facilitation Therapy along with Home care plan
Other: Nerve Flossing Technique — Tibial Nerve:
  1. Passively flex the hip while dorsiflexing and everting the ankle to create tension; flex the knee to unload, then extend and plantarflex to reload.
  2. Flex the hip, extend the knee, and dorsiflex and evert the ankle to induce tension; flex the hip to unload, then extend and plantarflex to reload.
  3. Lift the leg, flex the hip, and extend the knee; dorsiflex and evert the ankle to induce tension, then plantarflex to unload.
  Common Peroneal Nerve:
  1. Passively flex the hip and plantarflex and invert the ankle to induce tension; flex the knee to unload, then extend and dorsiflex to reload.
  2. Flex the hip, extend the knee, and plantarflex and invert the ankle to induce tension; flex the hip to unload, then extend and dorsiflex to reload.
  3. Lift the leg, flex the hip, and extend the knee; plantarflex and invert the ankle to induce tension, then dorsiflex to unload.
  Arms: Group B Nerve Flossing Technique along with Home care plan

SUMMARY:
The aim of this study is to determine the comparative effects of intraneural facilitation therapy and nerve flossing technique on pain, balance, gait, and quality of life in Diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Intraneural Facilitation Therapy is a novel manual therapy technique that seeks to enhance endoneurial capillary circulation, bias blood flow into the neural fascicle, and reverse intrafascicular ischemia. To redirect blood to the ischemic nerves, this passive approach involves tractioning skin, distending visceral tissues, stretching muscles, mobilizing joints, and stretching blood vessels. The Nerve Flossing Technique is an emerging treatment approach that aims to improve neurodynamic, range of motion, and quality of life. Intraneural Facilitation and Nerve Flossing Techniques address diabetic peripheral neuropathy, and their effectiveness in improving pain, balance, gait, and quality of life remains un-compared.

This randomized clinical trial will be conducted at Social Security Hospital, and Siddique Family Hospital, Gujranwala. 44 Participants who meet the inclusion criteria will be selected through a non-probability convenience sampling technique and randomly allocated into two groups using an online randomizer tool. Participants will be included in Groups A (Intraneural Facilitation Therapy) and Group B (Nerve Flossing Technique). A total of 24 sessions (3x/week for 8 weeks) will be conducted, lasting 60 minutes each.. A Numeric Pain Rating scale will be used to assess pain, the Berg Balance Scale (BBS) to assess balance, a 4-item Dynamic Gait Index to assess Gait, and the Quality of Life-Diabetic Neuropathy (QOL-DN) for quality of life. Assessment will be carried out at baseline (before treatment), after the 8th week (post-intervention), and at a 2-month follow-up. The data will be entered and analyzed using the IBM SPSS Statistics 27.0 version. Statistical significance will be set at p ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (diagnosed by the physician)
* Score >3 on Michigan Neuropathy Screening Instrument-Questionnaire and score >2 on MNSI-Physical Examination
* Diabetic peripheral neuropathy symptoms below the ankle (numbness, tingling, burning, sharp pain, increased sensitivity, etc.)

Exclusion Criteria:

* Presence of any other systemic disease rather than diabetes such as end-stage renal failure, uncontrolled hypertension, severe dyslipidemia, chronic liver disease, autoimmune disease, advanced chronic obstructive pulmonary disease, etc.
* Diabetic ulcer in either foot
* Total or partial amputation of lower extremities
* Active inflammations or other inflammatory neuropathies including chronic inflammatory demyelinating polyneuropathy, proximal diabetic neuropathy, chemotherapy-induced peripheral neuropathy, autonomic neuropathies, or other neuropathies not associated with DM such as B12 deficiency
* History of fracture, strain, history of trauma leading to nerve injuries in the last year.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 8 week
  Numeric Pain Rating Scale is a subjective measure 11 point (0-10) numerical scale which is a commonly used outcome measure to assess pain intensity, including in patients with diabetic peripheral neuropathy. Its score ranges from 0 indicating no pain at all to 10 indicating worst pain. In NPRS, 0 for No pain, 1-3 range for Mild pain, 4-6 range for Moderate pain, and 7-10 indicates Severe pain.
Michigan Neuropathy Screening Instrument | 8 week
  Michigan Neuropathy Screening Instrument (MNSI) is a simple, non-invasive, and valid tool for screening DPN in diabetic patients. The initial section of the assessment tool comprises a self-administered questionnaire (15 yes-or-no questions) focusing on foot sensation, including aspects like discomfort, numbness, and temperature sensitivity. The subsequent segment involves a brief physical examination such as visual inspection of the feet, testing ankle reflexes using a tendon hammer, assessing vibration perception utilizing a 128 Hz tuning fork, and evaluating tactile sensation through the application of a 10 gm Semmes-Weinstein Monofilament (SWM). A score greater than 3 on the MNSI-Q and greater than 2 on the MNSI-PE suggests diabetic peripheral neuropathy.
Quality of Life- Diabetic Neuropathy Questionnaire | 8 week
  The Norfolk QOL-DN is an extensive and validated 47-item questionnaire that has been developed to encompass the complete range of Diabetic Neuropathy (DN) symptoms associated with small fiber, large fiber, and autonomic neuropathy. It is composed of two sections: one focusing on the symptoms experienced by diabetic patients and the other on how the patient's neuropathy affects their activities of daily living (ADLs). The questionnaire items are divided into six different domains, namely overall quality of life, symptoms, ADLs, physical functioning/large fiber, small fiber, and autonomic neuropathy. The symptom domain (items 1-7) will allocated a score of 1 or 0, denoting the presence or absence of the specified symptoms. Apart from items 31 and 32, the remaining items were evaluated using a 5-point scale (0-4, ranging from "No Problem" to "Severe Problem").A score range of 2-9 classified the neuropathy as mild, 10-19 as moderate, and greater than or equal to 20 as severe.
BERG BALANCE SCALE | 8 week
  The BBS is a postural balance scale containing 14 items including standing and sitting unsupported, reaching forward, and placing the alternating foot on a stool. Administering the BBS takes approximately 15 min. Each of the 14 items is scored on a 5-level ordinal scale from 0 ("unable to perform or requiring help") to 4 ("normal performance"), thus providing a potential maximum score of 56 points.
4-Item Dynamic Gait Index | 8 week
  It is a shortened version of the Dynamic gait index. It consists of 4 items of Dynamic gait index such as horizontal head turns, vertical head turns, gait on level surfaces, and changes in gait speed. Each of the four items is scored on an ordinal scale from 0-3 with higher numbers indicating better performance of the specified task. Additionally, each item has specific criteria that must be met to be granted a specific score number. The test has a total score of 12.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Jabeen, MS-NMPT, Study Chair — Riphah International University
Locations (2):
- Pakistan (2):
  - Siddique Family Hospital, Gujranwala, Punjab Province
  - Social Security Hospital, Gujranwala, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Topp KS, Boyd BS. Structure and biomechanics of peripheral nerves: nerve responses to physical stresses and implications for physical therapist practice. Phys Ther. 2006 Jan;86(1):92-109. doi: 10.1093/ptj/86.1.92. PMID 16386065
- [Background] Intraneural Facilitation MR Bussell - US Patent App. 13/371,103, 2012
- [Background] Alnajafi KZ-S. The Impact of Intraneural Facilitation Therapy on Diabetic Peripheral Neuropathy Loma Linda University Electronic Theses, Dissertations & Projects 2021.
- [Background] BASUDEO RAJBHOR AG, SAURABH KUMAR. Comparison of Kinesio Taping and Nerve Flossing Technique on Balance, Gait and Ankle Flexibility in Diabetic Neuropathy. 2022.
- [Background] Dan Ran Castillo WJJ, Carvy Floyd Lucero, Mark Bussell, Ron Coleman, Karla Pieters, Jamie Hankins, Annette Boggs, Salem Dehom, Lorena Garcia, Ellen D'Errico, and Gayathri Nagaraj. A pilot study of intraneural facilitation versus standard physical therapy for prevention ofchemotherapy-induced peripheral neuropathy. Journal of Clinical Oncology. May31,2023.
- [Background] G.Tharani DJP, Dr. Jagatheesan Alagesan,Dr. Harikrishnan. N Exploring the Effectiveness of Peroneal Nerve Flossing in Alleviating Diabetic Peripheral Neuropathy Symptoms. Journal for Re Attach Therapy and Developmental Diversities. August6,2023
- [Background] Alshahrani A, Bussell M, Johnson E, Tsao B, Bahjri K. Effects of a Novel Therapeutic Intervention in Patients With Diabetic Peripheral Neuropathy. Arch Phys Med Rehabil. 2016 May;97(5):733-8. doi: 10.1016/j.apmr.2015.12.026. Epub 2016 Jan 22. PMID 26808781
- [Background] Goyat M, Saxena A, Goyal M. Study Protocol titled as "Effectiveness of neural mobilization in improving the ankle ROM and plantar pressure distribution in patients with diabetic peripheral neuropathy: A single group, pre post, quasi experimental study protocol". J Diabetes Metab Disord. 2022 Aug 15;21(2):2035-2041. doi: 10.1007/s40200-022-01106-z. eCollection 2022 Dec. PMID 36404825
- [Background] Sahba K, Berk L, Bussell M, Lohman E, Zamora F, Gharibvand L. Treating peripheral neuropathy in individuals with type 2 diabetes mellitus with intraneural facilitation: a single blind randomized control trial. J Int Med Res. 2022 Aug;50(8):3000605221109390. doi: 10.1177/03000605221109390. PMID 35922961
- [Background] Baker NA, Vuong D, Bussell M, Gharibvand L, Lee S, Tsao B. Prospective, Randomized, Double-Blinded, Sham-Controlled Pilot Study of Intraneural Facilitation as a Treatment for Carpal Tunnel Syndrome. Arch Rehabil Res Clin Transl. 2022 Mar 29;4(2):100193. doi: 10.1016/j.arrct.2022.100193. eCollection 2022 Jun. PMID 35756982